CLINICAL TRIAL: NCT03590327
Title: Transcranial Magnetic Stimulation for Apathy in Mild Cognitive Impairment
Acronym: TAMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Central Arkansas Veterans Healthcare System (U.S. Federal Agency); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2638-R; 1115904 (Other: Central Arkansas Veterans Healthcare System)
Record Dates: First submitted 2018-05-15; First posted 2018-07-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Apathy; Mild Cognitive Impairment; Transcranial Magnetic Stimulation; Loneliness; COVID; Neuropsychiatric Symptoms
MeSH Terms: conditions — Lethargy; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Apathy +, rTMS - (No Intervention): This arm will be followed without intervention
- rTMS (Active Comparator): This group will be randomized to receive rTMS treatment
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham (Sham Comparator): This group will be randomized to receive sham treatment
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — rTMS
  Arms: Sham; rTMS

SUMMARY:
Apathy, a profound loss of initiative and motivation, is often seen in older Veterans with memory problems. Apathy leads to serious health problems, increases dependency, and caregiver burden. If untreated, apathy hastens the progression to frank dementia. In a pilot study, the investigators found that apathy, working memory, and function can be restored using magnetic stimulation in some but not all older Veterans. The reason for this variation is unknown. The investigators propose a three-phase study in 125 older Veterans with mild memory problems. Their motivation, memory, and function will be measured periodically. Veterans with apathy that are eligible for treatment will receive either real or sham magnetic stimulation to the front part of their brain over 20 sessions. Genetic testing and biomarkers will be used to differentiate those who respond to magnetic stimulation from those who do not. Impact on function, quality of life, and rates of progression to dementia will also be studied.

A project modification was obtained to conduct a cross-sectional study, the COVID Dementia study. The cross-sectional study will examine the effect of the pandemic on MCI and AD patients and their caregivers ("individual COVID-related factors" such as, personally infected, death of a friend/family member, economic hardship, disruption in care, isolation), barriers to telehealth, caregiver distress, NPS, cognition (including onset of delirium), and function. Our goal is to develop a multi-pronged, remotely deliverable intervention to address consequences of healthcare disruptions in older Veterans with cognitive impairment.

Aim 1. To explore the association between COVID-related factors and neuropsychiatric symptoms in individuals with MCI and AD. Hypothesis: The number of COVID-related factors endorsed by caregivers will be positively correlated with the severity of NPI-Q in individuals with MCI and AD.

Aim 2. To assess cognition (telephonic version of the Montreal Cognitive Assessment; tMoCA12, and daily function (Functional Activities Questionnaire; FAQ13). Hypothesis: The number of COVID-related factors will be positively correlated with the severity of cognitive and functional deficits in individuals with MCI and AD.

Aim 3. To explore the associations among COVID-related factors and caregiver distress. Hypothesis: Caregiver resilience and perceived social support will modify the association between COVID-related factors and severity of distress in caregivers.

DETAILED DESCRIPTION:
Apathy, a profound loss of initiative and motivation, is often seen in older Veterans with memory problems. Apathy leads to serious health problems, increases dependency, and caregiver burden. If untreated, apathy hastens the progression to frank dementia. In a pilot study, the investigators found that apathy, working memory, and function can be restored using magnetic stimulation in some but not all older Veterans. The reason for this variation is unknown. The investigators propose a three-phase study in 125 older Veterans with mild cognitive impairment. Their motivation, other behavioral problems, memory, and function will be measured periodically. Veterans with apathy that are eligible for treatment will receive either real or sham magnetic stimulation to the dorsolateral prefrontal cortex over 20 daily sessions on consecutive week days. Genetic testing and biomarkers will be used to differentiate those who respond to magnetic stimulation from those who do not. Impact on function, quality of life, and rates of progression to dementia will also be studied.

A project modification was obtained to conduct a cross-sectional study, the COVID Dementia study. The cross-sectional study will examine the effect of the pandemic on MCI and AD patients and their caregivers ("individual COVID-related factors" such as, personally infected, death of a friend/family member, economic hardship, disruption in care, isolation), barriers to telehealth, caregiver distress, NPS, cognition (including onset of delirium), and function. Our goal is to develop a multi-pronged, remotely deliverable intervention to address consequences of healthcare disruptions in older Veterans with cognitive impairment.

Aim 1. To explore the association between COVID-related factors and neuropsychiatric symptoms in individuals with MCI and AD. Hypothesis: The number of COVID-related factors endorsed by caregivers will be positively correlated with the severity of NPI-Q in individuals with MCI and AD.

Aim 2. To assess cognition (telephonic version of the Montreal Cognitive Assessment; tMoCA12, and daily function (Functional Activities Questionnaire; FAQ13). Hypothesis: The number of COVID-related factors will be positively correlated with the severity of cognitive and functional deficits in individuals with MCI and AD.

Aim 3. To explore the associations among COVID-related factors and caregiver distress. Hypothesis: Caregiver resilience and perceived social support will modify the association between COVID-related factors and severity of distress in caregivers.

ELIGIBILITY:
Inclusion Criteria:

* meeting the modified Mayo Clinic criteria for MCI
* Having caregivers
* apathy threshold (NPI)
* MMSE 23
* On stable dose of antidepressants for at least a month (if applicable)

Exclusion Criteria:

PHASE I

* Uncontrolled diabetes mellitus (Fasting BS>200mg/dl, HbA1c>10)
* Renal disease requiring dialysis
* Uncontrolled blood pressure (>160/100, <100 systolic)
* Metastatic cancer or undergoing chemotherapy
* Deep venous thrombosis or myocardial infarction in past 3 months
* Uncontrolled malignant cardiac arrhythmia
* Cerebral aneurysm or intracranial bleed in past year
* Unstable angina in past month
* Unstable abdominal or thoracic aortic aneurysm (>4cm)
* End-stage congestive heart failure

EXCLUSIONARY DUE TO rTMS: ALL PHASE II AND SUBSET OF PHASE I THAT RECEIVE SINGLE SESSION rTMS

* Taking medications known to increase risk of seizures from 2012 Beers criteria such as bupropion, chlorpromazine, clozapine.
* Taking other medications known to increase risk of seizures such as tricyclic antidepressants.
* Taking ototoxic medications: Aminoglycosides, Cisplatin
* History of seizures/ seizures in first degree relatives
* Those with implanted device
* History of stroke, aneurysm, or cranial neurosurgery
* History of bipolar disorder
* Current alcohol related disorder needing medical treatment
* History of Tourette's syndrome or presence of motor tics
* History of abnormal electroencephalogram (EEG)

EXCLUSIONARY DUE TO CONFOUNDING WITH APATHY: PHASE II

* Current episode of Major Depressive Disorder
* Current use of stimulants
* Change in dose of dementia medications within 30 days
* Change in dose of antidepressants within 30 days

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Apathy Evaluation Scale Score | 2 weeks, 6 weeks, 6 months, 12 months, 24 months, 36 months, and 48 months
  Range 18-72 Lower score is improvement

SECONDARY OUTCOMES:
Change in Modified Mini Mental State Examination Score | 2 weeks, 6 weeks, 6 months, 12 months, 24 months, 36 months, and 48 months
  Range 0-100 Higher score is improvement
Change in Conner's Continuous Performance Test Commission Error percentage | 2 weeks, 6 weeks, 6 months, 12 months, 24 months, 36 months, and 48 months
  Range 0-100% Higher score is improvement

OTHER OUTCOMES:
Neuropsychiatric Inventory - Questionnaire | Through study completion, an average of 1 year
  To study the impact of COVID pandemic on neuropsychiatric symptoms of dementia. This outcome measure has questions pertaining to twelve neuropsychiatric symptoms seen in dementia. An aggregate score of the symptoms, caregiver distress and change during the COVID pandemic will be reported.
  Presence or lack of each domain is reported for this study. No range in score for this scale.
Functional Activities Questionnaire | Through study completion, an average of 1 year
  Measure of functional independence Range: 0-30 Higher score indicates higher dependence
UCLA Loneliness scale | Through study completion, an average of 1 year
  Measures loneliness Range 3-9 Higher score indicates higher loneliness
T-MoCA | Through study completion, an average of 1 year
  Measures global cognition Range: 0-22 Higher scores indicate better cognition

CONTACTS AND LOCATIONS:
Overall Officials: Prasad R. Padala, MBBS MBBS, Principal Investigator — Central Arkansas Veterans Healthcare System , Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma T, Padala PR, Mehta JL. Loneliness and Social Isolation: Determinants of Cardiovascular Outcomes. Curr Cardiol Rev. 2021;17(6):e051121190873. doi: 10.2174/1573403X17666210129101845. PMID 33511946
- [Background] Padala KP, Jendro AM, Wilson KB, Padala PR. Technology Use to Bridge the Gap of Social Distancing during COVID-19. J Geriatr Med Gerontol. 2020 Jun 29;6(2):10.23937/2469-5858/1510092. doi: 10.23937/2469-5858/1510092. No abstract available. PMID 33511321
- [Background] Padala KP, Parkes CM, Padala PR. Neuropsychological and Functional Impact of COVID-19 on Mild Cognitive Impairment. Am J Alzheimers Dis Other Demen. 2020 Jan-Dec;35:1533317520960875. doi: 10.1177/1533317520960875. PMID 32969235
- [Background] Padala PR, Boozer EM, Lensing SY, Parkes CM, Hunter CR, Dennis RA, Caceda R, Padala KP. Neuromodulation for Apathy in Alzheimer's Disease: A Double-Blind, Randomized, Sham-Controlled Pilot Study. J Alzheimers Dis. 2020;77(4):1483-1493. doi: 10.3233/JAD-200640. PMID 32925060
- [Background] Preston AM, Padala PR. Virtual reality on the verge of becoming a reality for geriatric research. Int Psychogeriatr. 2022 Feb;34(2):97-99. doi: 10.1017/S1041610221000867. Epub 2021 Jun 8. No abstract available. PMID 34099086
- [Background] Mintzer J, Lanctot KL, Scherer RW, Rosenberg PB, Herrmann N, van Dyck CH, Padala PR, Brawman-Mintzer O, Porsteinsson AP, Lerner AJ, Craft S, Levey AI, Burke W, Perin J, Shade D; ADMET 2 Research Group. Effect of Methylphenidate on Apathy in Patients With Alzheimer Disease: The ADMET 2 Randomized Clinical Trial. JAMA Neurol. 2021 Nov 1;78(11):1324-1332. doi: 10.1001/jamaneurol.2021.3356. PMID 34570180
- [Background] Mortby ME, Adler L, Aguera-Ortiz L, Bateman DR, Brodaty H, Cantillon M, Geda YE, Ismail Z, Lanctot KL, Marshall GA, Padala PR, Politis A, Rosenberg PB, Siarkos K, Sultzer DL, Theleritis C; ISTAART NPS PIA. Apathy as a Treatment Target in Alzheimer's Disease: Implications for Clinical Trials. Am J Geriatr Psychiatry. 2022 Feb;30(2):119-147. doi: 10.1016/j.jagp.2021.06.016. Epub 2021 Jul 1. PMID 34315645
- [Background] Okolichany R, Padala PR, Mooney S. Cognitive and Functional Abilities in an Older Adult Veteran Before and After Contracting COVID-19. J Alzheimers Dis Rep. 2022 Mar 25;6(1):115-120. doi: 10.3233/ADR-210055. eCollection 2022. PMID 35530116
- [Background] Preston AM, Brown L, Padala KP, Padala PR. Veterans Affairs Health Care Provider Perceptions of Virtual Reality: Brief Exploratory Survey. Interact J Med Res. 2022 Sep 2;11(2):e38490. doi: 10.2196/38490. PMID 36053568